CLINICAL TRIAL: NCT02598245
Title: Comparison of the Distance Between the Transobturator Tape (TOT) and the Urethra According to Two Different Placement Techniques of the Tape (TOT 8/4 vs TOT 6/3)
Brief Title: Comparison of TOT 8/4 Versus TOT 6/3
Acronym: URGE-III
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Klinikum der Universität Köln (Other)
Responsible Party: Principal Investigator, Professor Dr. Wolfram Jäger, Professor, Klinikum der Universität Köln
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 15-012
Record Dates: First submitted 2015-11-04; First posted 2015-11-05 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Urinary Incontinence
Keywords: urinary incontinence, CESA, VASA, TOT, TVT
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TOT 8/4 (Active Comparator): Transobturator sling (TOT) is placed according to the original description. Instead of a "Metzenbaum Scissor" which should guarantee the distance between the urethra and the sling a Hegar dilator sound of 4 mm diameter is used (Hegar 4). An additional Hegar dilator sound of 8 mm is placed in the urethra before tightening the sling and suturing the vaginal skin.
  Interventions: Device: TOT 8/4
- TOT 6/3 (Experimental): Transobturator sling (TOT) is placed according to the original description. Instead of a "Metzenbaum Scissor" which should guarantee the distance between the urethra and the sling a Hegar dilator sound of 3 mm diameter is used (Hegar 3). An additional Hegar dilator Sound of 6 mm is placed in the urethra before tightening the sling and suturing the vaginal skin.
  Interventions: Device: TOT 6/3

INTERVENTIONS:
Device: TOT 8/4 — placement of transobturator sling according to the TOT 8/4 technique
  Arms: TOT 8/4
Device: TOT 6/3 — placement of transobturator sling according to the TOT 6/3 technique
  Arms: TOT 6/3

SUMMARY:
Transobturator tapes (TOT) are placed according to the surgical technique described by Delorme et al. in patients with a previous cervico-sacropexy (CESA) or vagino-sacropexy (VASA). Before final Fixation of the tapes and suturing the vaginal skin a Hegar dilator sound with either 8 mm or 6 mm diameter is placed in the urethra and a second Hegar dilator sound with either 4 mm or 3 mm diameter is placed between the tape and the urethra. After suturing the vaginal skin the Hegar sounds are removed.

DETAILED DESCRIPTION:
Retrospective studies demonstrated that the distance between urethra and suburethral sling can vary considerably between 1 mm and 10 mm. In order to standardize the placement of the suburethral sling we choose two different distances between urethra and sling.

Transobturator tape (TOT) are placed according to the surgical technique described by Delorme et al. in patients with a previous cervico-sacropexy (CESA) or vagino-sacropexy (VASA). Before final fixation of the sling and suturing the vaginal skin a Hegar dilator sound with either 8 mm or 6 mm diameter is placed in the urethra and a second Hegar dilator sound with either 4 mm or 3 mm diameter is placed between the tape and the urethra. After suturing the vaginal skin the Hegar sounds are removed.

According to the used Hegar dilator sounds two different techniques are used:

TOT 8/4 or TOT 6/3.

ELIGIBILITY:
Inclusion Criteria:

* urinary incontinence

Exclusion Criteria:

* previous TOT or TVT

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Distance between urethra and transobturator sling | 2 weeks
  transvaginal ultrasound measurements

SECONDARY OUTCOMES:
Distance between urethra and transobturator sling | 16 weeks
  transvaginal ultrasound measurements

CONTACTS AND LOCATIONS:
Overall Officials: Wolfram Jager, Professor, Study Director — Head of the Department of Urogyne
Locations (1):
- Department of Obstetrics and Gynecology, University of Cologne, Cologne, North Rhine-Westphalia, Germany